CLINICAL TRIAL: NCT03509389
Title: The Prone XLIF. An Observational Pilot Study Based on Prospective Study
Brief Title: The Prone XLIF. A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: TheProneXLIF v.1-11/1/18
Record Dates: First submitted 2018-04-14; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Spinal Diseases
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational prospective study to evaluate the feasibility, effectiveness and the rate of complications of the XLIF (Extreme Lateral Interbody Fusion) performed in prone position to treat spinal diseases of the lumbar region.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients suffering from lumbar spinal disease that requires a circumferential fusion
* Patients suitable to undergo spinal fusion with an XLIF technique (according to the label indication/contraindications)
* Patients who are willing and able to provide written informed consent to surgery and study

Exclusion Criteria:

* a congenital or post-traumatic vertebral abnormality at the target level
* patients with a previous abdominal retroperitoneal surgery
* patients that refuses/not suitable to undergo a XLIF surgery in prone position
* subjects that are unable to provide a written informed consent to surgery and study
* subjects that are unable to will or intend
* pregnant women (declared before surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by a lumbar spinal disease, indicated for surgery requiring a lateral XLIF approach to the lumbar spine, eligible to perform the approach in a prone position.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-04-07 (Actual); Primary Completion 2019-04-07 (Estimated); Study Completion 2019-04-07 (Estimated)

PRIMARY OUTCOMES:
Complication rate | intraoperative
  Registration of intraoperative complications during surgery

SECONDARY OUTCOMES:
Oswestry Disability Index | in 5 days from surgery - 6 months follow-up
  Evaluation of clinical outcomes using Oswestry Disability Index (ODI) questionnaire. It is a scaled questionnaire from 0 to 100 in which the higher the value, the worst the outcome.
Length of surgery | intraoperative
  Evaluation of length of surgery
Subsidence rate | in 5 days from surgery
  Evaluation of subsidence rate at postoperative x-ray
Visual Analogic Score (VAS) leg and back | in 5 days from surgery - 6 months follow-up
  Evaluation of clinical outcomes using the VAS score, going from 0 to 10, where 0 means no pain and 10 the worst pain possible.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy